CLINICAL TRIAL: NCT04862767
Title: Multi-center, Open Label, Phase Ib Clinical Trial to Evaluate Safety, Tolerance and Efficacy of TASO(TGF-β2 Targeting Anti-sense Oligonucleotide)-001 in Combination With Recombinant Interleukin-2 in Advanced or Metastatic Solid Tumor
Brief Title: TASO-001 in Combination With Recombinant Interleukin-2(Aldesleukin) in Advanced or Metastatic Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Autotelicbio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ATB-301-001
Record Dates: First submitted 2021-03-17; First posted 2021-04-28 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Solid Tumor
Keywords: Autotelicbio; TASO; ATB-301; TGF-β2; Anti-sense Oligonucleotide; Interleukin-2; Aldesleukin
MeSH Terms: interventions — aldesleukin

STUDY DESIGN:
Intervention Model Description: 3+3 design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TASO-001 (Experimental): level 1 of TASO-001 in combination with recombinant IL-2(Aldesleukin)(3+3) next than level 2 or level -1 of TASO-001 in combination with recombinant IL-2(Aldesleukin)
  Interventions: Drug: TASO-001((TGF-β2 targeting anti-sense oligonucleotide); Combination Product: Aldesleukin

INTERVENTIONS:
Drug: TASO-001((TGF-β2 targeting anti-sense oligonucleotide) — 96 hour continuous infusion
Combination Product: Aldesleukin — SC, Bid

SUMMARY:
To evaluate safety, tolerance and efficacy of TASO(TGF-β2 targeting anti-sense oligonucleotide)-001 in combination with recombinant interleukin-2(Aldesleukin) in advanced or metastatic solid tumor and to find appropriate dose for phase 2 clinical trial.

DETAILED DESCRIPTION:
This clinical trial is conducted by dividing into two cohorts according to the dose of the test drug, starting with Cohort 1, and confirming whether DLT occurs until 14 days after the 2nd cycle of the test drug administration and proceed with Cohort 2 after discussion by DMC. Recruitment of each cohort is applied with a 3+3 design.

ELIGIBILITY:
Inclusion Criteria:

1. Adults over 19 years old on the day of consent
2. Pathologically confirmed solid cancer
3. Patients with advanced or metastatic solid timour failed or tolerable with standard therapy.
4. A person who has a tumor lesion that can safely undergo tissue biopsy during administration of the test drug and can provide tissues stored at the clinical trial agency or tissue obtained from a tissue biopsy conducted before the first administration of the test drug

Exclusion Criteria:

1. Those who have been treated with IL-2 or TGF-β inhibitors other than test drugs (e.g., anti-sense oligonucleotide, antibody, TGF-b receptor inhibitor)
2. Chemotherapy within 21 days or at least 5 half-lives (whichever is shorter) prior to first dose of study treatment.
3. Immunotherapy within 2 weeks prior to first dose of study treatment.
4. Major surgery within 4 weeks prior to first dose of study treatment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-08-21 (Actual)

PRIMARY OUTCOMES:
Incidence of MTD (Tolerability) | 4weeks(DLT)
  MTD and RP2D are determined

SECONDARY OUTCOMES:
ORR(objective response rate) | every 8 weeks, and up to 14 days after the last dose of TASO-001
  In case the best overall response expressed as CR or PR by RECIST v1.1 and iRECIST, the rate of subjects should be presented for each dose group.
DCR(Disease control rate) | every 8 weeks, and up to 14 days after the last dose of TASO-001
  In case the best overall response expressed as CR, PR or SD by RECIST v1.1 and iRECIST, the rate of subjects should be presented for each dose group.
DoR(Duration of response) | every 8 weeks, and up to 14 days after the last dose of TASO-001
  Median, standard deviation and 95% confidential interval of DoR is estimated by the Kaplan-Meier method.
PFS(Progression free survival) | every 8 weeks, up to 14 days after the last dose of TASO-001
  : Median, standard deviation and 95% confidential interval of PFS is estimated by the Kaplan-Meier method.
OS(Overall survival) | every 8 weeks, up to 14 days after the last dose of TASO-001
  : Median, standard deviation, 95% confidential interval of OS is estimated by Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: James Jun, M.D., Study Director — Autotelicbio
Locations (1):
- Seoul National University Hospital, Seoul, South Korea